CLINICAL TRIAL: NCT02809859
Title: CPAP In-home Assessment USA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA176
Record Dates: First submitted 2016-06-19; First posted 2016-06-22 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Investigational CPAP device (Experimental): Fisher & Paykel Healthcare CPAP Device
  Interventions: Device: Fisher & Paykel Healthcare CPAP Device

INTERVENTIONS:
Device: Fisher & Paykel Healthcare CPAP Device — Fisher & Paykel Healthcare CPAP Device

SUMMARY:
The study is to evaluate the product reliability, therapy effectiveness and user feedback of a Continuous Positive Airway Pressure (CPAP) device in-home for up to 6 months.

DETAILED DESCRIPTION:
Existing and Naïve CPAP users will be recruited into a 6 month in-home study Participants will attend 5 study visits at day 0, 7, 30, 60 and 180. Outcome of the clinical investigation include downloadable device data reports, device error reports and participants perception questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Aged 22 and over
* Diagnosed with Obstructive Sleep Apnea (OSA) and prescribed Positive Airway Pressure (either Continuous positive airway pressure (CPAP) or AutoCPAP)
* For experienced users of PAP (CPAP or AutoCPAP) - you must be using PAP of more than 4 hours/night for 70% during the last 30 days.

Exclusion Criteria:

* Contraindicated for PAP (CPAP or AutoCPAP) therapy
* Has other significant sleep disorders (e.g periodic leg movements, insomnia, central sleep apnea)
* Has obesity hypoventilation syndrome or congestive heart failure
* Requires supplemental oxygen with their PAP (CPAP or AutoCPAP) device
* Has implanted electronic medical devices (e.g cardiac pacemakers)
* Pregnant or think they may be pregnant
* Not fluent in spoken and written English.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2016-07; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matt Uhles, Principal Investigator — Clayton Sleep Institute
Locations (4):
- United States (4):
  - Alabama Sleep Clinic, Huntsville, Alabama
  - Pulmonary Disease Specialists - Central Florida Sleep Centre, Kissimmee, Florida
  - Clayton Sleep Institute, St Louis, Missouri
  - Ohio Sleep Medicine and Neurosciences Institute, Dublin, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Investigational CPAP Device
Started | 139
Completed | 125
Not Completed | 14

BASELINE CHARACTERISTICS:
Arm/Group | Investigational CPAP Device
Number analyzed (Participants) | 139
Age, Continuous [Mean (Full Range); unit: years] — Population: Age wasn't provided by one of the participants
  years
    number analyzed (Participants) | 138
    (all) | 55.5 [29 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 89
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Apnea Hypopnea Index (AHI), Measured as Number of Events/Hour.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: events/hr
Arm/Group | Investigational CPAP Device
Number analyzed (Participants) | 139
events/hr | 1.9 (2.9)

2. Primary Outcome: Log of Safety Related Events, Measured as Number of Participants That Experienced Unacceptable Safety Related Faults
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Investigational CPAP Device
Number analyzed (Participants) | 139
participants | 0

3. Primary Outcome: Machine Reported Faults, Measured as Number of Patients With Machine Faults
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Investigational CPAP Device
Number analyzed (Participants) | 139
participants | 3

4. Primary Outcome: Participant Reported Faults, Measured as Number of Participant Complaints
Time Frame: 6 months
Measure: Number; unit: complaints
Arm/Group | Investigational CPAP Device
Number analyzed (Participants) | 139
complaints | 9

5. Secondary Outcome: How Many Participants Slept Acceptably, Well or Very Well Throughout the Night on the CPAP Device
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Investigational CPAP Device
Number analyzed (Participants) | 139
participants | 134

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the study period of each participant (i.e. 6 months)
Arm/Group | Investigational CPAP Device
All-Cause Mortality (participants affected / at risk) | 1/139
Serious Adverse Events (participants affected / at risk) | 2/139
Other Adverse Events (participants affected / at risk) | 0/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational CPAP Device (N=139)
Community acquired pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Community acquired pneumonia assessed to be unrelated to trial
Atrial Fibrillation (Cardiac disorders) | 1 (1) — Atrial Fibrillation assessed to be unrelated to trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT02809859/Prot_SAP_000.pdf